CLINICAL TRIAL: NCT04641052
Title: Effects of Music Intervention on Pain, Anxiety and Vital Signs in Patients With Endoscopic Retrograde Cholangiopancreatography
Brief Title: The Effects Of Music In Endoscopic Retrograde Cholangiopancreatography Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Yeliz Ciğerci, Assistant Proffesor PhD, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020\481
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Endoscopic Retrograde Cholangio-Pancreatography; Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Intervention Group (Experimental): The music intervention group will be listened to the music by the researchers for the duration of 15 minutes before the procedure as well as the standard care.
  Interventions: Other: Music listening
- No Intervention Group (No Intervention): The control group patients will receive standard care only

INTERVENTIONS:
Other: Music listening — The music type will be chosen by the patients and researchers will not have any influence on their choices.
  Arms: Music Intervention Group

SUMMARY:
This study aims to investigate the effect of music listening on patients who will have Endoscopic Retrograde Cholangio-Pancreatography Procedure on vital signs, anxiety, and pain. This will be a randomized controlled experimental study.

The study will be conducted with two groups: the intervention group (n=35) and the control group (n=35). The control group will receive standard care while the intervention group, in addition to standard care, will be listened to music by the researchers for 15 minutes before the procedure.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 or above,
* with a scheduled ERCP procedure
* with the ASA grade level of I-II clinically
* without a hearing/speech impairment
* willing to participate in the research
* without a mental problem or diagnosis of psychiatric disorder
* without any a diagnosis of depression

Exclusion Criteria:

* Patients with an emergency ERCP procedure
* with a hearing/speech impairment
* not willing to participate in the research
* with a mental problem or diagnosis of psychiatric disorder
* with a diagnosis of depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale for Anxiety (VAS-A) | 1 Hour
  VAS-A is a 10 cm long measuring instrument with the score range from 0 to 10 with 0 points showing "no anxiety" and 10 points showing "I feel a lot of anxiety"
Visual Analog Scale for Pain (VAS) | 2 Hours
  VAS scale is a single-dimensional scale that is commonly used to evaluate pain severity. According to VAS, pain intensity is rated as "no pain" with 0 points, and "the most severe pain imaginable" with 10 points. Pain intensity ranges were determined by VAS as follows; mild pain below 3 points, as moderate pain between 3 and 6 points, and as severe pain above 6 points.The VAS pain scale was applied to the patients once on the first postoperative day, for the level of pain they felt.

SECONDARY OUTCOMES:
Vital Signs | 4 Hours
  The systolic and diastolic blood pressure will be measured with " MICROLIFE BP A 150 AFIB" device by the researchers.
Vital Signs | 4 hours
  Heart rate values of the patients will be measured with a finger type oximeter by the researchers.
Vital Signs | 4 hours
  SpO2 values of the patients will be measured with a finger type oximeter by the researchers.

CONTACTS AND LOCATIONS:
Overall Officials: Yeliz CIGERCI, Phd, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Sciences university Hospital, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No